CLINICAL TRIAL: NCT06989931
Title: A Clinical Study on the Safety and Effectiveness of Intracranial Distal Access Catheter in Neurointerventional Therapy
Brief Title: Intracranial Distal Access Catheter in Neurointerventional Therapy
Status: Completed | Type: Observational
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Collaborators: Tianjin Happy Life Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: STA-2023-01-0A
Record Dates: First submitted 2025-04-15; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke; Intracranial Aneurysms
MeSH Terms: conditions — Ischemic Stroke; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who using the Intracranial Distal Access Catheter to complete the procedure: Patients with mechanical thrombectomy for acute ischemic stroke, treatment of intracranial aneurysms and other ischemic and hemorrhagic diseases, requiring the use of Intracranial Distal Access Catheter to complete the procedure (such as poor vascular access conditions, lesions located in secondary or higher branches of cerebral vessels, inability of conventional guiding catheters in place and providing effective support. Treatment with Flow-divert devices, covered stents, etc.)
  Interventions: Device: Intracranial Distal Access Catheter

INTERVENTIONS:
Device: Intracranial Distal Access Catheter — Patients with mechanical thrombectomy for acute ischemic stroke, treatment of intracranial aneurysms and other ischemic and hemorrhagic diseases, requiring the use of Intracranial Distal Access Catheter(X-Track) to complete the procedure

SUMMARY:
The study objective is to evaluate the safety and effectiveness of Intracranial Distal Access Catheter in neurointerventional therapy.

DETAILED DESCRIPTION:
Patients with mechanical thrombectomy for acute ischemic stroke, treatment of intracranial aneurysms and other ischemic and hemorrhagic diseases, requiring the use of Intracranial Distal Access Catheter to complete the procedure were eligible. At last, 124 retrospective and prospective subjects in 6 centers were screened in this trial, and 114 subjects were successfully enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18-80 years old.
* Patients with mechanical thrombectomy for acute ischemic stroke, treatment of intracranial aneurysms and other ischemic and hemorrhagic diseases, requiring the use of Intracranial Distal Access Catheter to complete the procedure (such as poor vascular access conditions, lesions located in secondary or higher branches of cerebral vessels, inability of conventional guiding catheters in place and providing effective support. Treatment with Flow-divert devices, covered stents, stent grafts, etc.)
* Patients agree to participate in the study and sign the informed consent form.（only prospective enrolled patients)

Exclusion Criteria:

* Intracranial Distal Access Catheter is used during the interventional therapy of non-neurovascular diseases, such as peripheral vascular and coronary artery diseases.
* Interventional procedure is performed with other distal catheters or devices with the same function before using Intracranial Distal Access Catheter.

Ordinary guiding catheters can be used to establish access to complete the procedure without the use of Intracranial Distal Access Catheter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mechanical thrombectomy for acute ischemic stroke, treatment of intracranial aneurysms and other ischemic and hemorrhagic diseases, requiring the use of Intracranial Distal Access Catheter to complete the procedure (such as poor vascular access conditions, lesions located in secondary or higher branches of cerebral vessels, inability of conventional guiding catheters in place and providing effective support. Treatment with Flow-divert devices, covered stents, stent grafts, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Technical success rate | immediately after procedure
  It is defined as the proportion of subjects where Intracranial Distal Access Catheter can reach the expected position to successfully deliver the device and meet the treatment needs.
  Special note: If the patient uses more than one Intracranial Distal Access Catheters during the procedure, as long as any Intracranial Distal Access Catheter is delivered successfully, the patient is considered to achieve successful delivery with Intracranial Distal Access Catheter.
  Technical success rate (%) = number of patients successfully delivered/number of patients analyzed * 100%

SECONDARY OUTCOMES:
Catheter delivery success rate | immediately after procedure
  It is defined as the proportion of Intracranial Distal Access Catheter where Intracranial Distal Access Catheter can reach the expected position to successfully deliver the device and meet the treatment needs.
  Special note: If the patient uses more than one Intracranial Distal Access Catheters during the procedure, the statistics are based on whether the delivery of each Intracranial Distal Access Catheter is successful or not.
  Catheter delivery success rate (%) = number of successful catheter delivery/total number of catheters used * 100%
Incidence of device-related adverse events | from the procedure to patients discharged from the hospital, anticipated average 5 days
Incidence of device-related serious adverse events | from the procedure to patients discharged from the hospital, anticipated average 5 days

OTHER OUTCOMES:
Device operation performance (device compatibility) | intra-procedure
  The evaluation of device compatibility is to evaluate whether it can be compatible with other devices(such as Coils, Flow-divert devices, Stenosis stents, Thrombectomy Stents ) The evaluation criteria for device compatibility is
  * Yes
  * No
Device operation performance (supporting capability) | intra-procedure
  The evaluation criteria for supporting capacity are as follows:
  * Excellent: During the delivery of therapeutic devices, the Intracranial Distal Access does not withdraw..
  * Good: During the delivery of therapeutic devices, the Intracranial Distal Access Catheter withdraws slightly, but the adjustment has no significant impact on the procedure.
  * Poor: During the delivery of therapeutic devices, the Intracranial Distal Access Catheter withdraws seriously, requiring repeated adjustments to significantly prolong the procedure time.
Device operation performance (pushing resistance) | intra-procedure
  The evaluation criteria for pushing resistance are as follows:
  * Excellent: Smooth push
  * Good: Slight resistance but not affecting use
  * Poor: Large resistance, affecting the proper placement and use

CONTACTS AND LOCATIONS:
Overall Officials: JUN DONG, Associate chief physician, Principal Investigator — Rizhao People's Hospital
Locations (6):
- China (6):
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Jiangmen Xinhui District People's Hospital, Jiangmen, Guangdong
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The Sixth People's Hospital of Nantong, Nantong, Jiangsu
  - People's Hospital of Rizhao, Rizhao, Shandong
  - The Affiliated Hospital of Yunnan University, Kunming, Yunnan